CLINICAL TRIAL: NCT06966934
Title: The Application of Nasopharyngeal Airway Combined With Nasal High-flow Oxygen Therapy During Painless Gastroscopy in Patients With Obesity
Brief Title: Nasopharyngeal Airway Combined With Nasal High-flow Oxygen Therapy During Painless Gastroscopy in Obesity Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20250327-10
Record Dates: First submitted 2025-04-25; First posted 2025-05-13 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-04

CONDITIONS: Hypoxia; Obesity; Gastrostomy
Keywords: Obese patients; sedative gastroscopy; high-flow nasal oxygen therapy
MeSH Terms: conditions — Hypoxia; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HFNC30L/min (No Intervention): The patient receives pre-oxygenation with pure oxygen at 30 L/min for 1 minute. After sedation, when the patient's breathing becomes slightly slower but stable and the eyelash reflex disappears, continue to supply oxygen at a flow rate of 30 L/min
- HFNC30L/min AND NPA (Experimental): The patient receives pre-oxygenation with pure oxygen at 30 L/min for 1 minute. After sedation, the nasopharyngeal airway (NPA) is inserted when the patient's breathing becomes slightly slow but stable and the eyelash reflex disappears
  Interventions: Device: NPA

INTERVENTIONS:
Device: NPA — After sedation, the nasopharyngeal airway (NPA) is inserted when the patient's breathing becomes slightly slow but stable and the eyelash reflex disappears.
  Arms: HFNC30L/min AND NPA

SUMMARY:
Gastroscopy is a commonly used, direct, and reliable method for screening and diagnosing digestive tract diseases. However, as an invasive examination, it can cause adverse reactions such as pain, nausea, vomiting, and choking cough in patients. Compared with ordinary gastroscopy, painless gastroscopy offers higher comfort and satisfaction for patients and greater convenience for endoscopists during operation.

The most common complication of painless gastroscopy diagnosis and treatment is hypoxia. High-flow nasal cannulala (HFNC) provides a higher oxygen concentration and flow rate than an ordinary nasal catheter. It has the functions of heating and humidifying, which can relieve the pressure on the nasal mucosa cilia, keep the airway unobstructed and moist, and reduce the risk of epistaxis. Due to changes in airway anatomical structures such as fat accumulation in the head and neck and hyperplasia of oropharyngeal soft tissues, obese patients are more prone to hypoxia during gastroscopy under sedation. Therefore, HFNC is often used to reduce the occurrence of hypoxia.

The nasopharyngeal airway (NPA) is used to maintain the patency of the upper respiratory tract and is suitable for patients with spontaneous breathing but partial obstruction of the upper respiratory tract. It is worth exploring how effective the combination of HFNC and NPA is in improving hypoxemia in obese patients during sedation.

DETAILED DESCRIPTION:
Gastroscopy is a commonly used, direct, and reliable method for screening and diagnosing digestive tract diseases. However, as an invasive examination, it can cause adverse reactions such as pain, nausea, vomiting, and choking cough in patients. With the promotion of comfortable medical technology, more patients choose painless gastroscopy. Compared with ordinary gastroscopy, patients have a higher level of comfort and satisfaction, and it is more convenient for endoscopists to operate. Obesity is a chronic and multisystemic disease, and its prevalence is on the rise worldwide. It is estimated that by 2035, the prevalence of obesity will increase from 14% of the world's population to 24% in 2035. Due to the relationship between obesity and obesity-related comorbidities (such as dyslipidemia, hypertension, diabetes, cardiovascular diseases, and even certain types of cancer), it is necessary and important to actively control and treat obesity. Therefore, it is strongly recommended that such people undergo gastroscopy, whether it is for preoperative examination of bariatric surgery or for the diagnosis and treatment of gastrointestinal diseases. With the increase in the number of obese patients, the proportion of the patient group undergoing sedated gastrointestinal endoscopy has also increased. During painless gastroscopy, respiratory depression has always been one of the common adverse reactions. The incidence of hypoxia in obese patients during sedated gastroscopy is higher than that in patients with normal body weight, and it increases with the increase of the body mass index. Therefore, high-flow nasal cannulala (HFNC) is often used clinically to reduce the occurrence of hypoxia in obese patients during painless gastroscopy.

HFNC is a new type of ventilation method. It can provide patients with a high flow rate (20-70L/min) of oxygen through a special nasal cannula, and the oxygen concentration can be adjusted (21%-100%). It has the functions of heating and humidifying, which can relieve the pressure on the nasal mucosa cilia, keep the airway unobstructed and moist, and reduce the risk of epistaxis. In addition, HFNC can generate positive airway pressure (3-7cmH2O), increase the end-expiratory volume, help with alveolar re-expansion, prevent atelectasis, and reduce shunt. Obese patients have fat accumulation in the head and neck, hyperplasia of oropharyngeal soft tissues, reduced lung compliance, reduced lung volume and functional residual capacity. Some obese patients also suffer from obstructive sleep apnea, which increases the risk of hypoxemia in obese patients .

The Nasopharyngeal Airway (NPA) is a commonly used ventilation assistance tool. It is a soft and curved tube that is inserted through the nasal cavity so that the front end of the tube is located in the pharynx, bypassing the parts where obstruction may occur (such as the backward displacement of the tongue root, etc.), thus establishing a gas passage to allow air to smoothly pass through the upper respiratory tract into the trachea and lungs, ensuring the normal ventilation of patients. It is suitable for patients with spontaneous breathing but partial obstruction of the upper respiratory tract. For obese patients, NPA has significant advantages in reducing airway obstruction, being easy to insert, having good tolerance, not affecting oral cavity operations, reducing respiratory resistance, and reducing complications. It is an effective tool for managing the airway of obese patients. Therefore, the investigators propose the hypothesis that the use of NPA combined with HFNC during painless gastroscopy in obese patients can further reduce the incidence of hypoxia in obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing painless gastroscopy;
2. Patients with an age greater than 18 years old;
3. American Society of Anesthesiologists (ASA) physical status classification from Grade I to Grade III;
4. Body Mass Index (BMI) greater than 28 kg/m²

Exclusion Criteria:

1. Patients with contraindications to endoscopic procedures or those who refuse sedation/anesthesia;
2. Patients allergic to propofol, eggs, soybeans, milk, etc.;
3. Patients with gastrointestinal tract obstruction and gastric emptying disorders;
4. Patients with acute pharyngitis, tonsillitis, and upper respiratory tract infections;
5. Patients in the acute exacerbation stage of respiratory diseases such as asthma, bronchitis, and chronic obstructive pulmonary disease (COPD);
6. Patients with acute arrhythmia and those with severe heart diseases (congenital diseases, valvular diseases);
7. Patients with severe hepatic and renal insufficiency who require alternative treatment;
8. Patients with severe mental disorders who need medications to control their symptoms;
9. Patients with moderate or above anemia, abnormal coagulation function, and hematological diseases;
10. Patients with nasal cavity lesions leading to severe nasal congestion;
11. Pregnant and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
incidence of hypoxia | 6 mintues after gastroscopy completion
  75% ≤ SpO2 < 90% for <60 s

SECONDARY OUTCOMES:
incidence of subclinical respiratory depression | 6 mintues after gastroscopy completion
  90% ≤ SpO2 < 95%
incidence of severe hypoxia | 6 mintues after gastroscopy completion
  SpO2 < 75% for any duration or 75% ≤ SpO2 < 90% for ≥60 s
periprocedural complications | 6 mintues after gastroscopy completion
  vomit and nausea
airway associated complications | 6 mintues after gastroscopy completion
  incidence of patients with glossoptosis, excessive oropharynx secretion, laryngeal spasm,bronchospam
adverse event | 6 mintues after gastroscopy completion
  patients dispalyed unpredicatable movement, overexcitement and delirium after sedation with propofol
airway intervention to handle hypoxia | 6 mintues after gastroscopy completion
  jaw lift,increase the flow of oxygen, Mask ventilation,Intubation

CONTACTS AND LOCATIONS:
Overall Officials: Lihai Chen, Doctor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No